CLINICAL TRIAL: NCT02238223
Title: Post Marketing Surveillance of Alesion® (Epinastine Hydrochloride) Tablet
Brief Title: Postmarketing Surveillance to Investigate the Safety and Efficacy Information of Alesion® Tablet
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 262.290
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients without experience in treatment with epinastine
  Interventions: Drug: Alesion®

INTERVENTIONS:
Drug: Alesion®

SUMMARY:
Study to investigate the safety and efficacy information of Alesion® Tablet under the proper use in daily clinical practice after new treatment guideline for allergic rhinitis, bronchial asthma, eczema, dermatitis, urticaria, pruritus, prurigo and psoriasis vulgaris with itching

ELIGIBILITY:
Inclusion Criteria:

All the patients who:

* haven't treatment experience of epinastine product;
* have at least one out of following diseases. allergic rhinitis, eczema, dermatitis, pruritus, prurigo, urticaria, psoriasis with itching, bronchial asthma

Exclusion Criteria:

* Alesion® Tablet is contraindicated for the patients with history of hypersensitivity to any ingredients of Alesion® Tablet in package insert. However, it is unknown whether a patient is hypersensitive to the ingredients of the product in almost cases. And this survey is drug utilization study to observe actual use in any patients. Therefore exclusion criteria is not set in the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients without experience treating of epinastine are selected by physicians at medical institutions
Sampling Method: Non-Probability Sample
Enrollment: 2001 (Actual)
Dates: Start 2004-04; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | up to 24 months
  classified by Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of adverse drug reactions classified by patient's background/treatment factors | up to 24 months

SECONDARY OUTCOMES:
Overall assessment of efficacy by investigator on a 3-point scale | after 24 months